CLINICAL TRIAL: NCT00593944
Title: A Phase 1, Open-Label, Multiple-Dose, Dose-Escalation Study of MDX-1342 in Patients With CD19-Positive Refractory/Relapsed Chronic Lymphocytic Leukemia
Brief Title: Study of MDX-1342 in Patients With Chronic Lymphocytic Leukemia (CLL)
Acronym: MDX1342-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1342-02; IM130-002 (Other: BMS)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Chronic Lymphocytic Leukemia; B cell; leukemia; lymphocyte; antibody; monoclonal; cancer; blood
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Neoplasms | interventions — MDX-1342 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will receive active MDX-1342.
  Interventions: Biological: MDX-1342

INTERVENTIONS:
Biological: MDX-1342 — MDX-1342 is given as a 90 minute i.v. infusion. Patients will receive one of the following dose levels, 0.7, 7, 40, 200, 1000, 2000 mg/dose.

SUMMARY:
The purpose of this study is to see at what dose MDX-1342, a monoclonal antibody, is safe and tolerable for patients with chronic lymphocytic leukemia (CLL). Information on any responses that patients may have to the drug will also be collected.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is a monoclonal hematopoietic disorder characterized by a progressive expansions of lymphocytes of B-cell lineage. These small, mature-appearing lymphocytes accumulate in the blood, bone marrow, lymph nodes, and spleen. CLL is a common leukemia in the wester world and accounts for 25% to 30% of adult leukemias. CD19,an integral membrane protein, is expressed by pro-B cells and functions as a co-stimulatory molecule that regulates mature B-cell activation and enhances B-cell proliferation. MDX-1342, a fully human monoclonal antibody, has demonstrated to specifically bind to human CD19 antigen with high affinity. Therefore, it is theorized that MDX-1342 will block activation of B cell stimulation, decreasing the number of cancerous B cell clones.

ELIGIBILITY:
Inclusion Criteria:

* relapsed/refractory CD19-positive CLL
* At least 28 days since prior treatment for CLL
* ECOG PS 0-2
* Screening laboratory values must be met

Exclusion Criteria:

* No prior anti-CD19 antibody tx
* No active, uncontrolled infection
* No prior allogeneic bone marrow transplant
* No autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
incidence and severity of treatment-emergent adverse events | all events will be followed to resolution

SECONDARY OUTCOMES:
response | 12 weeks
clinical laboratory tests | study duratation - each visit
physical examination | study duration - each visit
electrocardiogram | at screening and study completion
diagnostic testing | at screening and study completion
pharmacokinetics sampling | at each dosing visit

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Oncology Consultants, PA, Houston, Texas